CLINICAL TRIAL: NCT03886909
Title: The Effects of a Prehabilitation Exercise Program in Adults Receiving a Hematopoietic Stem Cell Transplant
Brief Title: Impact of Prehabilitation in Oncology Via Exercise- Bone Marrow Transplant
Acronym: IMPROVE-BMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Shin Mineishi, Professor, Public Health Science, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010914
Record Dates: First submitted 2019-03-12; First posted 2019-03-22 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Hematopoietic Stem Cell Transplant; Hematologic Diseases; Physical Activity; Prehabilitation
Keywords: Exercise; Hematopoietic Stem Cell Transplant; Physical function; Quality of Life
MeSH Terms: conditions — Hematologic Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-Based Prehabilitation (Active Comparator): Will be offered an individual one-on-one appointment for an exercise introduction session with an exercise and cancer specialist and periodical phone calls to support and adapt the exercise program. The exercises should be done home-based for 5 times a week until the time of transplant.
  Interventions: Behavioral: Exercise
- Prehabilitation Education (Active Comparator): Will be offered a prehabilitation and stem cell education class at the Penn State Hershey Cancer Institute.
  Interventions: Behavioral: Prehabilitation Education

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention is at least 2 weeks lasting (till the day transplant is taking place) 5-times weekly resistance training intervention combined with aerobic exercise (mostly walking).
  Arms: Home-Based Prehabilitation
Behavioral: Prehabilitation Education — Participant will receive a prehabilitation and stem cell education class which will be held at the Penn State Cancer Institute.
  Arms: Prehabilitation Education

SUMMARY:
The purpose of this study is to determine whether patients are able to participate in a prehabilitation program (prior to the beginning of treatment) which includes: (1) a home-based exercise program or (2) just a prehabilitation education session.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplant may have the potential for severe side effects, including functional (reduced aerobic capacity, reduced muscle strength) and psychosocial (e.g. reduced quality of life, increased fatigue) detriments.

Evidence shows that exercise is considered to be an effective treatment approach in hematopoietic stem cell transplant patients during and after treatment with regard to the above mentioned side-effects. Also, prehabilitative exercise in colon and lung cancer patients was shown as feasible and effective. However, no experience exists with regard to prehabilitation exercise in hematopoietic stem cell transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Hematological cancer (e.g. Acute Myeloid Leukemia, Chronic Lymphocytic Leukemia, Multiple Myeloma, Non-Hodgkin Lymphoma, etc.)
* Hematological cancer in remission
* Females and males ≥18 years of age
* Fluent in written and spoken English
* Must be able to provide and understand informed consent
* Must have an ECOG score of ≤ 2
* Scheduled for an inpatient autologous or allogeneic stem cell transplant at Penn State Cancer Institute
* ≥ 2 weeks until scheduled transplant
* Primary attending physician approval

Exclusion Criteria:

* Hematological cancer not in remission
* Evidence in the medical record of an absolute contraindication (e.g. Heart insufficiency > NYHA III or uncertain arrhythmia; uncontrolled hypertension; reduced standing or walking ability) for exercise
* Any other comorbidities or musculoskeletal complications that preclude participation in the exercise programs as deemed by the exercise interventionist
* Uncontrolled hypertension
* Receiving non-transplant related chemotherapy and/or radiotherapy
* Not fluent in written and spoken English
* Active infections, hemorrhages, and cytopenias that could place transplant patients at risk for further adverse events, deemed by the exercise interventionist, physician and/or nurse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of the exercise intervention: 50% of included patients actually complete at least one third of the exercise sessions | Through study completion, an average of 18 months
  The exercise intervention will be considered feasible if 50% of included patients actually complete at least one third of the exercise sessions prescribed for 2 weeks or more.
Acceptability of the exercise intervention: more than 50% of the patients approached | During recruitment
  The exercise intervention will be considered acceptable if more than 50% of the patients approached agree to receive at least the first exercise session.
Safety of the exercise intervention: questionnaire | Through the study completion, an average of 18 months
  Within the questionnaire we will assess whether musculoskeletal occur (yes/no; ongoing; location; severity (mild-life threatening); daily activities affected). The intervention will be considered as safe if less than 25% of included patients report mild musculoskeletal impairments and less than 5% experienced musculoskeletal injuries (defined as symptoms lasting a week or longer and or requiring the attention of a medical professional).

SECONDARY OUTCOMES:
Health-related Quality of Life: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30, version 3.0) | Through study completion, an average of 18 months
  QoL will be assessed with the validated 30-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30, version 3.0).
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Bone Marrow Transplant-related Quality of Life: EORTC QLQ-HDC29 | Through study completion, an average of 18 months
  Quality of Life will be assessed with the validated 29-item self-assessment questionnaire of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire- High Dose Chemotherapy- 29 Items (EORTC QLQ-HDC29).
  The QLQ HDC29 module includes 29 items, consisting of six multi-item scales and eight single-items. For the multi-item scales and single-item scales a high score is equivalent to worse or more symptoms/problems.
Fatigue | Through study completion, an average of 18 months
  Fatigue will be assessed with the Multidimensional Fatigue Inventory (MFI) which is a 20-item, multidimensional self-assessment questionnaire.
  Respondents use a scale ranging from 1 to 7 to indicate how aptly certain statements regarding fatigue represent their experiences. Higher total scores correspond with more acute levels of fatigue.
Sleep | Through study completion, an average of 18 months
  Sleep quality and sleep problems will be assessed with the validated and frequently used Pittsburgh Sleep Quality Index (PSQI).
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Depression | Through study completion, an average of 18 months
  Depressive symptoms will be assessed with the 20-item Center for Epidemiological Studies Depression Scale (CES-D).
  Zero for 'Rarely', 1 for 'Some or a little of the time', 2 for 'Occasionally or a moderate amount of time', 3 for 'Most or all of the time'. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Short Questionnaire to Assess Health-Enhancing Physical Activity | Through study completion, an average of 18 months
  Physical activity behavior in the domains of commuting activity, leisure time activities such as cycling, walking, and sports, household and occupational activity will be assessed via a standardized and validated questionnaire, the Short QUestionnaire to ASsess Health-enhancing Physical Activity (SQUASH).
  Household work and activities at work or school were prestructured for intensity. A basic intensity score of 2 and 5 for light and intense activities, respectively. Total minutes of activity are calculated for each question by multiplying frequency (days/week) by duration (min/day). Activity scores for separate questions are calculated by multiplying total minutes of activity by the intensity score. The total activity score is calculated by taking the sum of the activity scores for separate questions. Higher values equals more time spent completing the activity.
Godin Physical Activity Questionnaire | Through study completion, an average of 18 months
  Physical activity behavior in the domains of commuting activity, leisure time activities such as cycling, walking, and sports, household and occupational activity will be assessed via a standardized and validated questionnaire, the Godin Physical Activity Questionnaire.
  Total weekly leisure activity is calculated in arbitrary units by summing the products of the separate components, as shown in the following formula:
  Weekly leisure activity score = (9 × Strenuous) + (5 × Moderate) + (3 × Light) Higher activity score = more active
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events | Through study completion, an average of 18 months
  Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) will be used to collect information on severity and interference of symptoms and adverse events.
Body Pain: Brief Pain Inventory- Short form | Through study completion, an average of 18 months
  Bodily pain will be assessed using the Brief Pain Inventory- Short form (BPI-SF).
  The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The pain interference score corresponds to the item on pain interference. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Physical Function: Short Physical Performance Battery | Through study completion, an average of 18 months
  Objectively-measured physical function will be assessed using the Short Physical Performance Battery (SPPB).
  The SPPB is an accumulation of balance tests, 4-meter gait speed, and 5-chair stands. Based on the time needed to complete the chair stands, a score is given. A summation of scores from all tests is taken, ranging from 0 -12. A higher score = Higher physical function.
Aerobic Capacity: Six Minute Walk Test | Through study completion, an average of 18 months
  Objectively-measured physical function will be assessed using the Six Minute Walk Test (6MWT).
  Distance walked during 6 minutes (measured in meters) is measured. Longer distance = higher aerobic capacity.
Physical Function: Timed-Up-and-Go Test | Through study completion, an average of 18 months
  Objectively-measured physical function will be assessed using the Timed-Up-and-Go test (TUG).
  Time taken to stand up from a chair, walk 10 meters around an obstacle, and return to seated position is measured in seconds. Lower time = better physical function.
Fall Risk | Through study completion, an average of 18 months
  Functional balance will be assessed using the Berg Balance Scale.
  Scoring: A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Score is summation of all items. Highest Total Score = 56 Interpretation: 0-20: Wheelchair bound; 21-40: Walking with assistance; 41-56: Independent

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — Penn State College of Medicine, Hershey
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potiaumpai M, Schmitz KH, Mineishi S, Naik S, Wirk B, Rakszawski K, Ehmann WC, Claxton D, Nickolich M, Zemel BS, Zheng H. IMPROVE-BMT: a protocol for a pilot randomised controlled trial of prehabilitation exercise for adult haematopoietic stem cell transplant recipients. BMJ Open. 2023 Jan 18;13(1):e066841. doi: 10.1136/bmjopen-2022-066841. PMID 36657760